CLINICAL TRIAL: NCT01583088
Title: Can Diaphragm Pacing Delay Non Invasive Ventilation in Amyotrophic Lateral Sclerosis ? a Randomized Controlled Study
Brief Title: Early Stage Amyotrophic Lateral Sclerosis Phrenic Stimulation
Acronym: RespiStimALS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: in the absence of benefits and because of a statistically significant excess mortality in the group of patients receiving active stimulation.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: ARSla (Association pour la recherche sur la SLA) (Unknown); Fondation Thierry Latran (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AOM11046
Record Dates: First submitted 2012-04-20; First posted 2012-04-23 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-04

CONDITIONS: Amyotrophic Lateral Sclerosis; Respiratory Insufficiency
Keywords: Amyotrophic lateral sclerosis,; Diaphragm; Mechanical ventilation; Phrenic nerve stimulation; Respiratory insufficiency
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- phenic nerve stimulation (Experimental): effective phenic nerve stimulation NeurX™ (Synapse Biomedical)
  Interventions: Device: phenique nerve stimulation NeurX™ (Synapse Biomedical)
- sham (Sham Comparator): sham phenic nerve stimulation
  Interventions: Device: sham phrenic nerve stimulation

INTERVENTIONS:
Device: phenique nerve stimulation NeurX™ (Synapse Biomedical) — phenique nerve stimulation NeurX™ (Synapse Biomedical)
  Arms: phenic nerve stimulation
Device: sham phrenic nerve stimulation — sham phenic nerve stimulation
  Other Names: sham phenic nerve stimulation
  Arms: sham

SUMMARY:
ALS is is characterized by a progressive degeneration of motor neurons, leading to progressive weakness of muscles, including respiratory muscles, the diaphragm. Although specific therapy is lacking, correct respiratory therapy improves quality of life and increases survival. Substituting the failing respiratory muscles by non invasive mechanical ventilatory assistance (NIV) is the current standard of care. Intradiaphragmatic phrenic nerve stimulation is a new treatment and has been the object of a preliminary international proof-of-concept multicenter trial. This trial suggests that the intradiaphragmatic phrenic nerve stimulation slows down the rate of decline of the diaphragm. Our new hypothesis is that phrenic stimulation induces diaphragm conditioning and can delay the need for mechanical ventilation in ALS patients. We will study, during 24 months, 2 groups of 37 patients at the beginning of the respiratory dysfunction, using a intradiaphragmatic phrenic nerve stimulation in one group and a sham stimulation in the other group. Although, all the patients will be implanted, thus, at the end of the study, all the patients will receive effective stimulation.

DETAILED DESCRIPTION:
ALS is is characterized by a progressive degeneration of upper and lower motor neurons, leading to progressive weakness of bulbar, limb, thoracic and abdominal muscles. Although specific therapy is lacking, correct respiratory therapy improves quality of life and increases survival. Substituting the failing respiratory muscles by non invasive mechanical ventilatory assistance (NIV) is the current standard of care.Intradiaphragmatic phrenic nerve stimulation, has been the object of a preliminary proof-of-concept multicenter trial (ClinicalTrials.gov NCT00420719).

Aim of the study : To test the hypothesis that phrenic stimulation induced diaphragm conditioning can delay the need for mechanical ventilation in ALS patients.

Methods : It is a double blind randomized study. Patients presenting with early signs of respiratory impairment (VC between 85 and 60%), but with a preserved electromyographic response of the diaphragm to phrenic nerve stimulation, will be randomized in 2 groups. All the patients will be treated according to current standards of care. They will all be implanted with a phrenic stimulator, and then randomized between actual diaphragm conditioning and sham stimulation.

Respiratory function will be followed up on a trimonthly basis, with polysomnography and diaphragmatic EMG biannually. NIV (+ stimulation for both groups), will be initiated according to currently recommended criteria of hypoventilation.

The main outcome of the study will be the number of months between the phrenic nerve implantation and the introduction of NIV. Currently available data, showing that diaphragm pacing can increase the number of patients without NIV at 2 years from 2,5% to 15% of the patients, requires the enrollment of 37 patients in each group. Secondary end-points will include i.Survival ii. Effects on sleep iii. Quality of life and daily activities

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis is laboratory-supported probable, probable, or definite according to the World Federation of Neurology El Escorial criteria
* Forced Vital Capacity (FVC) from 80 - 60% of predicted values at enrollment
* Bilateral phrenic nerve function acceptable as demonstrated by bilateral diaphragm EMG recordings and nerve conduction times without axonal lesion

Exclusion Criteria:

* Active cardiovascular disease that would increase the risk of general anesthesia. (FEVG<60%)
* Underlying pulmonary diseases that were present prior to ALS that would effect pulmonary tests independent of ALS, in particular COPD with FEV1<30%
* Pre-existing implanted electrical device such as a pacemaker or cardiac defibrillator
* respiratory infection or decompensation in the last 30 days
* Marked obesity affecting suitability for surgery
* Significant scoliosis or chest deformity affecting suitability for surgery
* Pre-existing diaphragm abnormality such as a hiatal hernia or paraesophageal hernia
* Patient on NIV, CPAP or Oxygen for a reason other than ALS
* Criteria for NIV (VC<50% of predicted values and/or Pi max and SNIP<60% of predicted values; and/or nocturnal desaturations without SAOS and/or PaCO2>45 mm d'Hg)
* Supine VC<50% of predicted values

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Survival without NIV 2 years after the phrenic nerve implantation. | 2 years

SECONDARY OUTCOMES:
global survival from onset disease | 2 years
effects on sleep | 24 months
Quality of life and daily activities | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalez-Bermejo Jesus, Md, PhD, Principal Investigator — APHP
Locations (1):
- APHP, GH Pitié Salpêtrière, Paris, France

REFERENCES:
- [Derived] Guimaraes-Costa R, Similowski T, Rivals I, Morelot-Panzini C, Nierat MC, Bui MT, Akbar D, Straus C, Romero NB, Michel PP, Menegaux F, Salachas F, Gonzalez-Bermejo J, Bruneteau G; RespiStimALS team; contributors to the RespiStimALS study were:. Human diaphragm atrophy in amyotrophic lateral sclerosis is not predicted by routine respiratory measures. Eur Respir J. 2019 Feb 14;53(2):1801749. doi: 10.1183/13993003.01749-2018. Print 2019 Feb. PMID 30523161
- [Derived] Gonzalez-Bermejo J, Morelot-Panzini C, Tanguy ML, Meininger V, Pradat PF, Lenglet T, Bruneteau G, Forestier NL, Couratier P, Guy N, Desnuelle C, Prigent H, Perrin C, Attali V, Fargeot C, Nierat MC, Royer C, Menegaux F, Salachas F, Similowski T. Early diaphragm pacing in patients with amyotrophic lateral sclerosis (RespiStimALS): a randomised controlled triple-blind trial. Lancet Neurol. 2016 Nov;15(12):1217-1227. doi: 10.1016/S1474-4422(16)30233-2. Epub 2016 Oct 11. PMID 27751553